CLINICAL TRIAL: NCT01797991
Title: Étude Pilote DEXEL-RH: Comparaison de Deux schémas Posologiques de DEXaméthasone en prévention Des Réactions d'Hypersensibilité au paclitaXEL
Brief Title: Comparison of Two Regimens of Dexamethasone in the Prevention of Hypersensitivity Reactions to Paclitaxel, a Pilot Study
Acronym: DEXEL-RH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CE12.270
Record Dates: First submitted 2013-02-19; First posted 2013-02-25 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Prevention of Hypersensitivity Reactions to Paclitaxel
Keywords: Hypersensitivity, drug
MeSH Terms: conditions — Drug Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (dexamethasone per os) (Active Comparator): * Dexamethasone 20 mg per os 12 hours and 6 hours before paclitaxel (form: opaque white capsules)
  * Matching placebo for dexamethasone IV (NaCl 0,9%) 30 minutes before paclitaxel
  Interventions: Drug: Dexamethasone per os; Drug: Matching placebo for dexamethasone IV
- Group B (dexamethasone IV) (Experimental): * Dexamethasone 20 mg IV 30 minutes before paclitaxel
  * Matching placebo for dexamethasone per os (lactose capsule) 12 hours and 6 hours before paclitaxel (form: opaque white capsules)
  Interventions: Drug: Dexamethasone IV; Drug: Matching placebo for dexamethasone per os

INTERVENTIONS:
Drug: Dexamethasone per os
  Arms: Group A (dexamethasone per os)
Drug: Matching placebo for dexamethasone IV
  Arms: Group A (dexamethasone per os)
Drug: Dexamethasone IV
  Arms: Group B (dexamethasone IV)
Drug: Matching placebo for dexamethasone per os
  Arms: Group B (dexamethasone IV)

SUMMARY:
This is a prospective, randomized, unicentric, two-arm, parallel, controlled, and double blind pilot study.

The purpose of this pilot study is to assess the feasibility of a trial designed to compare the quality of life of patients taking dexamethasone in two different ways to prevent hypersensitivity reactions to paclitaxel.

Dexamethasone given intravenously (IV) 30 minutes before paclitaxel could improve quality of life, could adequately prevent hypersensitivity reactions to paclitaxel and could reduce adverse effects compared to dexamethasone given orally 12 hours and 6 hours before paclitaxel.

DETAILED DESCRIPTION:
Primary objective:

To assess the feasibility of a randomized, parallel, two-arm, controlled and double blind trial designed to compare the quality of life of patients taking dexamethasone 20 mg IV 30 minutes before paclitaxel with those taking a standard dose of dexamethasone, 20 mg orally 12 hours and 6 hours before paclitaxel, in patients taking paclitaxel every two to three weeks for a minimum of two cycles in order to estimate a sample size.

Secondary objectives:

Between the two study groups, to compare:

* Quality of life during the first two cycles of chemotherapy;
* Efficacy of dexamethasone in preventing acute hypersensitivity reactions to paclitaxel in the first two cycles of chemotherapy;
* Adverse effects associated with dexamethasone on a daily basis during the first seven days of the first two cycles of chemotherapy.

Eligible patients will be randomized in a 1:1 ratio to one of the two study groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated at the outpatient clinic or admitted to the oncology unit of Notre-Dame Hospital between February 4, 2013 and July 19, 2013;
* Patient diagnosed with cancer;
* Patient starting a chemotherapy containing paclitaxel every two to three weeks for a minimum of two cycles;
* Patient aged 18 years and over;
* Patient able to give free and informed consent and who agrees to participate by signing the consent form;
* Patient able to complete the questionnaire on quality of life EORTC QLQ-C30 and the personal logbook.

Exclusion Criteria:

* Patient unable to speak English or French;
* Patient who has previously received paclitaxel;
* Patient receiving a prescription of paclitaxel bound to albumin;
* Patient is currently under treatment with systemic corticosteroids or has received systemic corticosteroids during the last week;
* Patient in another research protocol evaluating a different chemotherapy regimen;
* Patient who had an allergic reaction to taxanes;
* Patient with severe intolerance to lactose;
* Patient with an allergy or a severe intolerance to products containing castor oil (eg.: cyclosporine and vitamin K).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Quality of life assessed by the self-administered quality of life core questionnaire (QLQ-C30) version 3.0 from the European Organisation for Research and Treatment in Cancer (EORTC) | Day before chemotherapy (Day 0) of the first cycle of chemotherapy
  Comparison of the scores according to the EORTC Scoring Manual.
Quality of life assessed by the self-administered questionnaire QLQ-C30 version 3.0 from the EORTC | Day 6 of the first cycle of chemotherapy
  Comparison of the scores according to the EORTC Scoring Manual.
Quality of life assessed by the self-administered questionnaire QLQ-C30 version 3.0 from the EORTC | Day before chemotherapy (Day 0) of the second cycle of chemotherapy
  Comparison of the scores according to the EORTC Scoring Manual.
Quality of life assessed by the self-administered questionnaire QLQ-C30 version 3.0 from the EORTC | Day 6 of the second cycle of chemotherapy
  Comparison of the scores according to the EORTC Scoring Manual.

SECONDARY OUTCOMES:
Acute hypersensitivity reactions assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03 | During the administration of paclitaxel (Day 1) of the first cycle of chemotherapy
  Proportion of participants that had acute hypersensitivity reactions. Adverse events selected: allergic reaction, anaphylaxis, dyspnea, chest pain, hypertension, back pain and abdominal pain.
Acute hypersensitivity reactions assessed by the NCI CTCAE version 4.03 | During the administration of paclitaxel (Day 1) of the second cycle of chemotherapy
  Proportion of participants that had acute hypersensitivity reactions. Adverse events selected: allergic reaction, anaphylaxis, dyspnea, chest pain, hypertension, back pain and abdominal pain.
Use of rescue medication | During the administration of paclitaxel (Day 1) of the first cycle of chemotherapy
  Proportion of participants that needed rescue medication
Use of rescue medication | During the administration of paclitaxel (Day 1) of the second cycle of chemotherapy
  Proportion of participants that needed rescue medication
Adverse effects self-assessed by a personal logbook | Assessed on a daily basis from Day 1 to Day 7 of the first cycle of chemotherapy
  Proportion of participants with adverse effects
Adverse effects self-assessed by a personal logbook | Assessed on a daily basis from Day 1 to Day 7 of the second cycle of chemotherapy
  Proportion of participants with adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Samouelian, M.D., Ph. D., Principal Investigator — CHUM
Locations (1):
- Oncology oupatient clinic and oncology unit; CHUM Notre-Dame Hospital, Montreal, Quebec, Canada